CLINICAL TRIAL: NCT05022537
Title: Clinical Outcomes of Percutaneous Nephrolithotomy Following Retrograde Percutaneous Nephrostomy Access Using Novel Device in Comparison to Antegrade Access
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nadeem N Dhanani, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-20-1269
Record Dates: First submitted 2021-08-19; First posted 2021-08-26 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Kidney Stone
Keywords: nephrostomy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (retrograde nephrostomy) (Experimental)
  Interventions: Device: retrograde nephrostomy
- Control Group ( antegrade nephrostomy) (Active Comparator)
  Interventions: Device: antegrade nephrostomy

INTERVENTIONS:
Device: retrograde nephrostomy — this will consist of one visit to a urologist for retrograde nephrostomy placement using a Retroperc device with lithotomy performed in the same visit and follow up at 4 weeks and 6 months.
  Arms: Treatment (retrograde nephrostomy)
Device: antegrade nephrostomy — this will consist of two visits, first to the interventional radiologist for antegrade nephrostomy placement followed by another visit to the urologist for lithotomy with follow up at 4 weeks and 6 months
  Arms: Control Group ( antegrade nephrostomy)

SUMMARY:
The purpose of this study is to compare relevant clinical outcomes in patients requiring percutaneous nephrostomy for urolithiasis treatment between those who undergo an antegrade approach versus a retrograde approach and to determine which clinical characteristics predict success of lithotomy with anterograde or retrograde percutaneous nephrostomy approaches.

ELIGIBILITY:
Inclusion Criteria:

-Renal pelvis and proximal ureteral stones >10 mm confirmed with non-contrast computed tomography

Exclusion Criteria:

* Suspected pyelonephritis.
* Prior percutaneous nephrolithotomy procedure in affected kidney.
* Mid-ureteral or distal ureteral stones.
* Pregnancy.
* Anatomical abnormal kidney, including:

  * Horseshoe
  * Ectopic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy as measured by the time taken from diagnosis to nephrostomy access | end of procedure (about 4-8 weeks from diagnosis)
Treatment efficacy as measured by total time of access operation. | end of procedure( about 90 minutes after start of procedure)
Treatment efficacy as measured by total time of access operation fluoroscopy | end of procedure( about 90 minutes after start of procedure)
Treatment efficacy as measured by total time of lithotomy operation | end of procedure(about 3 hours after start of procedure)
Treatment efficacy as measured by total time of lithotomy operation fluoroscopy | (end of procedure)about 3 hours after start of procedure
Treatment efficacy as measured by length of post-operative hospital stay | 24 hours after procedure
Number of patients that are stone free | 6-12 weeks after procedure
  stone free is defined as <2mm on non-contrast computed tomography
Number of patients with symptom free survival as defined as lack of flank pain | 6-12 weeks after procedure
Number of patients with symptom free survival as defined as lack of presence of urinary or gastrointestinal symptoms, | 6-12 weeks after procedure
Number of patients with symptom free survival as defined as lack of limitations to work | 6-12 weeks after procedure
Number of patients with symptom free survival as defined as lack of limitations to social or daily activities. | 6-12 weeks after procedure

SECONDARY OUTCOMES:
Number of patients with nephrostomy access adequate for stone treatment | end of procedure( abut 3 hours from start of procedure)
Number of patients with normal vital signs | end of procedure( abut 3 hours from start of procedure)
Number of patients with normal laboratory values | 24 hours after procedure
  laboratory values include complete metabolic panel and urinalysis
Number of patients with an infection rate which is defined as a positive culture within the study time period | 6-12 weeks after procedure
Number of patients that require pain medication (defined as discharge with an opioid prescription). | 6-12 weeks after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem N Dhanani, MD,MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No